CLINICAL TRIAL: NCT00163163
Title: Carotid Atorvastatin Study In Hyperlipidemic Post-Menopausal Women: A Randomized Evaluation of Atorvastatin, Versus Placebo (CASHMERE)
Brief Title: Carotid Atorvastatin Study in Hyperlipidemic Post-Menopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A2581051
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Hypercholesterolaemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Blood Specimen Collection

INTERVENTIONS:
Procedure: Echographic measurements
Procedure: Blood samples

SUMMARY:
To evaluate the effect of atorvastatin 80 mg, versus placebo, given for 12 months on carotid intima-media thickness in postmenopausal women with moderate hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women defined as having Age =< 70 years with documented menopause
* Fasting LDL cholesterol 130 mg/ dl (3.37 mmol/l)and =< 190 mg/ dl (4.92 mmol/l) after 6 weeks of diet
* Triglycerides =< 4 g/l(4.52 mmol/l)
* Informed, written consent

Exclusion Criteria:

* Age > 70 years
* Unconfirmed menopause
* Overall duration of treatment with any HMG-CoA Reductase inhibitor > 3 months within the last year
* Patient treated with any lipid-lowering drugs within the last 6 weeks preceding the randomization
* History of myocardial infarction, coronary bypass surgery, angioplasty, stroke or TIA
* CPK levels > 3 times upper limit of normal
* Body Mass Index >= 30

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2003-01; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Mean change in carotid IMT from baseline to month 12.

SECONDARY OUTCOMES:
Mean change from baseline to month 12 of carotid internal diameter (ID)
wall cross sectional area (WCSA); carotid arterial mass (AM)
pulse pressure (PP); cross sectional distensibility and compliance (DC and CC)
pulse wave velocity (PWV); Lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (58):
- Belgium (10):
  - Pfizer Investigational Site, Afsnee GENT
  - Pfizer Investigational Site, Assenede
  - Pfizer Investigational Site, Brussels
  - Pfizer Investigational Site, Ertvelde
  - Pfizer Investigational Site, Ghent
  - Pfizer Investigational Site, Linkebeek
  - Pfizer Investigational Site, Sint-Niklaas
  - Pfizer Investigational Site, Tielt
  - Pfizer Investigational Site, Wetteren
  - Pfizer Investigational Site, Wondelgem
- France (45):
  - Pfizer Investigational Site, Achenheim
  - Pfizer Investigational Site, Ancerville
  - Pfizer Investigational Site, Augny
  - Pfizer Investigational Site, Bar-le-Duc
  - Pfizer Investigational Site, Bois-Colombes
  - Pfizer Investigational Site, Boissy-Saint-Léger
  - Pfizer Investigational Site, Bouzonville
  - Pfizer Investigational Site, Bœrsch
  - Pfizer Investigational Site, Colombey-les-Belles
  - Pfizer Investigational Site, Dammarie-les-Lys
  - Pfizer Investigational Site, Docelles
  - Pfizer Investigational Site, Dourdan
  - Pfizer Investigational Site, Eckbolsheim
  - Pfizer Investigational Site, Epinay S/orge
  - Pfizer Investigational Site, Étampes
  - Pfizer Investigational Site, Frouard
  - Pfizer Investigational Site, Gambsheim
  - Pfizer Investigational Site, Haguenau
  - Pfizer Investigational Site, Kilstett
  - Pfizer Investigational Site, Laxou
  - Pfizer Investigational Site, Le Grand-Quevilly
  - Pfizer Investigational Site, Le Mesnil-Esnard
  - Pfizer Investigational Site, Leuville-sur-Orge
  - Pfizer Investigational Site, Lingolsheim
  - Pfizer Investigational Site, Longpont-sur-Orge
  - Pfizer Investigational Site, Mars-la-Tour
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Moûtiers
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pont-à-Mousson
  - Pfizer Investigational Site, Pulnoy
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Saint-Max
  - Pfizer Investigational Site, Sainte-Geneviève-des-Bois
  - Pfizer Investigational Site, Sauvigny
  - Pfizer Investigational Site, Savigny-sur-Orge
  - Pfizer Investigational Site, Sotteville-lès-Rouen
  - Pfizer Investigational Site, Souffelweyersheim
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Terville
  - Pfizer Investigational Site, Toul
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Verdun
  - Pfizer Investigational Site, Vincennes
- Netherlands (3):
  - Pfizer Investigational Site, ED Voerendaal
  - Pfizer Investigational Site, EN Vaals
  - Pfizer Investigational Site, VE Maastricht

REFERENCES:
- [Derived] Gompel A, Boutouyrie P, Joannides R, Christin-Maitre S, Kearny-Schwartz A, Kunz K, Laurent S, Boivin JM, Pannier B, Pornel B, Struijker-Boudier HA, Thuillez C, Van Bortel L, Zannad F, Pithois-Merli I, Jaillon P, Simon T. Association of menopause and hormone replacement therapy with large artery remodeling. Fertil Steril. 2011 Dec;96(6):1445-50. doi: 10.1016/j.fertnstert.2011.09.010. Epub 2011 Oct 6. PMID 21982290
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2581051&StudyName=Carotid%20Atorvastatin%20Study%20in%20Hyperlipidemic%20Post-Menopausal%20Women